CLINICAL TRIAL: NCT02059967
Title: A Phase I Image-Guided Adaptive Radiotherapy Study Using Active Breathing Control (ABC) and Simultaneous Integrated Boost for Patients With Inoperable Non-Small Cell Lung Cancer
Brief Title: Phase I IGART Study Using Active Breathing Control and Simultaneous Boost for Patients With NSCLC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to no accrual.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13-09209; HM20000101 (Other: IRB); MCC-20000101 (Other: VCU Massey Cancer Center); NCI-2014-00163 (Registry Identifier: NCI)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Adenocarcinoma of the Lung; Large Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
Keywords: Lung
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Taxes; Carboplatin; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (IGART using ABC, SIVAB, paclitaxel, carboplatin) (Experimental): Patients undergo IGART using ABC 5 days a week for 7 weeks, for a total of 33 fractions with SIVAB during fractions 26-33. Patients also receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes once a week for 6 weeks.
  Interventions: Drug: Paclitaxel; Radiation: image-guided adaptive radiation therapy; Drug: carboplatin

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: 5beta,20-epoxy-1,2alpha,4,7beta,10beta, 6,12b-bis(acetyloxy)-12-(benzoyloxy)-1a,33,4,-4, Anzatax, Asotax, Bristaxol, Praxel, TAX, Taxol, Taxol Konzentrat
Radiation: image-guided adaptive radiation therapy — Undergo IGART
  Other Names: IGART, image-guided adaptive radiotherapy
Drug: carboplatin — Given IV
  Other Names: Blastocarb, Carboplat, Carboplatin Hexal, Carboplatino, Carbosin, Carbosol, Carbotec, CBDCA,; Novoplatinum, Paraplat, Paraplatin, Paraplatin AQ, Paraplatine, platinum, Ribocarbo

SUMMARY:
This phase I trial studies the side effects and best dose of image-guided adaptive radiation therapy using active breathing control when given together with chemotherapy and simultaneous integrated boost in treating patients with stage IIA-IIIB non-small cell lung cancer that cannot be removed by surgery. Image-guided adaptive radiation therapy aims radiation therapy right at the tumor so that higher radiation doses can be given without causing bad side effects. Giving these higher doses may help control the tumor better. Breathing causes organs and tissues, including the tumor, to move within the chest. Active breathing control may reduce the volume that needs to be treated. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving image-guided adaptive radiation therapy using active breathing control with chemotherapy and simultaneous integrated boost may be an effective treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of IGART.

Patients undergo IGART using active breathing control (ABC) 5 days a week for 7 weeks, for a total of 33 fractions with simultaneous integrated volume adapted boost (SIVAB) during fractions 26-33. Patients also receive paclitaxel intravenously (IV) over 1 hour and carboplatin IV over 30 minutes once a week for 6 weeks.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven (by biopsy or cytology), unresectable or inoperable lung cancer of the following histologic types: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, non-small cell carcinoma not otherwise specified.
* The tumor stage must be Stage IIA-IIIB (AJCC 7th edition). See http://aboutcancer.com/AJCC 7th lung 1.gif and http://aboutcancer.com/AJCC 7th lung 2.gif for staging.
* All detectable tumor must be encompassed by radiation therapy fields.
* 18-fluorodeoxyglucose PET is required for staging and treatment planning.
* Atelectasis, if present, must involve less than a complete lung.
* Laboratory values:

  * Neutrophils >1500/µL
  * Platelets >100,000/µL
  * Bilirubin < 1.5 mg/dL
  * Aspartate aminotransferase (AST; formerly serum glutamic oxaloacetic transaminase [SGOT]) < 2x upper limit normal
  * Alanine aminotransferase (ALT; formerly serum glutamic pyruvic transaminase [SGPT]) < 2x upper limit normal
  * Serum creatinine < 2.0 mg/dL
  * Glomerular filtration rate (GFR) calculated (kidney function test) within 30 days must be ≥ 59 mL/min
  * Pulmonary function test (PFT) with FEV-1 ≥ 1.0 L/sec
* Plan of curative radiotherapy with or without concurrent chemotherapy.
* Karnofsky Performance Scale score of ≥ 70%.
* Age ≥ 18 years old.
* Measurable disease on the planning CT.
* Patient must have a completed IMRT plan to 66 Gy in 2 Gy fractions with ≥ 95% of the PTV covered by the prescription dose, and the attending physician must have reviewed and approved the DVHs as follows:

  * total lung V20 Gy ≤ 30%
  * mean esophageal dose ≤ 34 Gy
  * esophageal planning organs-at-risk volume (PRV) V60 Gy ≤ 30%
  * heart V40 Gy ≤ 50%
  * maximum brachial plexus dose ≤ 66 Gy
  * maximum spinal cord PRV dose ≤ 50 Gy
  * maximum aorta dose ≤ 66 Gy
  * maximum main bronchus dose ≤ 66 Gy
  * maximum dose ≥ 66 Gy allowed in only one lobar bronchus.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Complete tumor resection, recurrent disease, or those patients eligible for definitive surgery.
* Prior radiation therapy to the thorax.
* Previous chemotherapy or previous biologic response modifiers for current lung cancer or within the past 5 years.
* Clinically significant pleural effusions, pericardial effusions, or superior vena cava syndrome.
* Oxygen supplementation required during therapy.
* Involvement of the brachial plexus, or infiltration of the aorta, heart, or esophagus.
* Tumors that affect more than one lobar bronchus, except the second involved bronchus in the right middle lobe bronchus.
* Unable to perform the BH procedures, unless tumor motion is ≤ 3 mm.
* Myocardial infarction within the last 6 months, symptomatic heart disease, uncompensated chronic obstructive pulmonary disease (COPD), or uncontrolled bronchospasms.
* History of a prior malignancy from which the patient has not been disease free for a minimum of 2 years, other than adequately treated basal/squamous skin cancer or in situ cervix cancer or other in situ malignancy.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the highest dose level at which =< 3 out of 7 patients experience a dose-limiting toxicity | 3 months
  (using daily image-guidance, deformable image registration, adaptive replanning at defined time points, and dose intensification at normal tissue tolerance) of radiotherapy delivered concomitantly with standard chemotherapy.

SECONDARY OUTCOMES:
Incidence of acute toxicity measured using the National Cancer Institution Common Terminology for Adverse Events version 4.0 | Up to 90 days from radiation therapy start
  Toxicities associated with higher dose per fraction during the SIVAB phase of the protocol will be tabulated and analyzed with respect to treatment dose, respective normal tissue structure and dose-volume parameters.
Incidence of late toxicity measured using the Radiation Therapy Oncology Group Late Radiation Morbidity Scoring | Up to 5 years
  Toxicities associated with higher dose per fraction during the SIVAB phase of the protocol will be tabulated and analyzed with respect to treatment dose, respective normal tissue structure and dose-volume parameters.
Practicability of the approach | Up to 5 years
  Variations in respiratory patterns, tumor and CTV positions, as well as tumor volumes will be assessed on the respective under-treatment imaging studies. The feasibility of deformable image registration will be benchmarked against manual contours of targets and normal tissue. The practicability of IGART will be measured by assessing the necessary time, IT and personnel resources needed to conduct the study.
Tumor response evaluated according to Response Evaluation Criteria in Solid Tumors v1.1 | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Weiss, MD, Principal Investigator — Virginia Commonwealth University